CLINICAL TRIAL: NCT07363226
Title: Efficacy of Two Different Exercises Approach: Core Stabilization Exercises Versus Traditional Rehabilitation on Adolescent Idiopathic Scoliosis-A Single Blind Randomized Control Trial
Brief Title: Effect of Core Stabilization Exercises Versus Traditional Rehabilitation in Adolescent With Idiopathic Scoliosis
Acronym: AIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Hind Khalid Ali AlQhtani, Principal investigator (physiotherapist), Armed Forces Hospitals, Southern Region, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: study-001
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Adolescence Idiopathic Scoliosis; Core Stabilization Exercise; Traditional Rehabilitation; Adolescents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stabilization exercises group (Experimental): A supervised core stabilization exercise program targeting deep and global trunk musculature including the transversus abdominis, multifidus, pelvic floor, diaphragm, rectus abdominis, erector spinae, and oblique muscles. The program was delivered three times per week for 12 weeks, with each session lasting 45 minutes. Exercises were progressively advanced from static to dynamic tasks according to participant tolerance and performance.
  Interventions: Behavioral: Core stabilization Exercises program
- Traditional Rehabilitation Exercise Program (Experimental): A supervised traditional physiotherapy program including postural correction exercises, diaphragmatic breathing, spinal mobility exercises, stretching of muscles on the concave side of the curve, and general strengthening exercises for trunk, pelvic, and shoulder girdle musculature. The program was delivered three times per week for 12 weeks, with each session lasting 45 minutes.
  Interventions: Behavioral: Traditional Rehabilitation exercises program

INTERVENTIONS:
Behavioral: Core stabilization Exercises program — A supervised core stabilization exercise program targeting deep and global trunk musculature including the transversus abdominis, multifidus, pelvic floor, diaphragm, rectus abdominis, erector spinae, and oblique muscles. The program was delivered three times per week for 12 weeks, with each session lasting 45 minutes. Exercises were progressively advanced from static to dynamic tasks according to participant tolerance and performance.
  Arms: core stabilization exercises group
Behavioral: Traditional Rehabilitation exercises program — Conventional Rehabilitation exercises commonly used in clinical practice for adolescents with idiopathic scoliosis
  Arms: Traditional Rehabilitation Exercise Program

SUMMARY:
This study aims to compare the effectiveness of core stabilization exercises versus traditional rehabilitation exercises in adolescents with idiopathic scoliosis. Participants are assigned to one of two intervention groups: a core stabilization exercise program or a traditional rehabilitation program. The study evaluates the impact of both interventions on spinal stability, posture, and functional outcomes. The results of this study may help identify more effective rehabilitation approaches for managing adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents aged 11-18 years
* Diagnosed with idiopathic scoliosis
* Cobb's angle between 10° and 40°
* Referred to physiotherapy

Exclusion Criteria:

* Congenital, neuromuscular, or secondary scoliosis
* Previous spine surgery or spinal correction
* Presence of rheumatologic, renal, cardiovascular, pulmonary, or vestibular disorders
* Inability to follow verbal instructions

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants who are biological Female
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cobb's Angle | Baseline and 12 weeks
  Cobb's angle measured using the DIERS Formetric 4D spinal analysis system in static mode

SECONDARY OUTCOMES:
1. Maximum Axial Vertebral Rotation (Max AVR) | Baseline and 12 weeks
  Measured using DIERS Formetric 4D
Pelvic Obliquity | Baseline and 12 weeks
  Measured using DIERS Formetric 4D
Quality of Life (QoL) | Baseline and 12 weeks
  The SRS-22 questionnaire consists of 22 items scored from 1 to 5, with total scores ranging from 1 (worst outcome) to 5 (best outcome). Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Hospital Southern Region, Khamis Mushait, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No